CLINICAL TRIAL: NCT02200679
Title: Study on Approach and Standards for Diagnosis, Prevention and Control of Autism Spectrum Disorder in Children in China
Brief Title: National Study on Autism Spectrum Disorder in China
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Principal Investigator, Yi Wang, Vice Prsident Chlidren's Hospital of Fudan University, Fudan University
Other Study IDs: 201302002
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism spectrum disorders; Prevalence; Diagnosis; Screen; Risk Factor; SRS; ASRS
MeSH Terms: conditions — Autism Spectrum Disorder; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood 2*5ml, (isolate Plasma, Serum and white cell) Hair, Urine(biosample will be collected only for Cases 1200 +Controls 1200)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Autism Spectrum Disorders: Cases were children living in target communities who are identified as positive based on questionnaire screen and the following diagnosis with DSM-Ⅳ, ADOS and ADI-R

SUMMARY:
The aims of the national population-based study on Autism Spectrum Disorder (ASD) include: (1) to understand the overall prevalence of ASD in children aged 6-12 years in 8 cities (n=120,000), (2) to explore environmental and genetic risk factors associated with ASD

DETAILED DESCRIPTION:
The study is a multicenter, cross-sectional study involing eight cities. The program includes a prevalence study and a risk factors analysis.

1. Prevalence study on ASD To estimate the national prevalence of ASD in Chinese pediatric population aged 6-12 years.

   1.1. Target population This 4-year study is initiated in the year of 2013 in eight cities of China . For each city, 3 communities with different economic levels were chosen including all children born within Jan 2001 to Dec 2007 (ages 6-12 years at screening) with local residency or have lived in the community over 6 months. The ASD children who are attending special education schools and meet with the inclusion criteria will also be included in the prevalence estimation.

   1.2. Sample size Based on the previous regional studies , we plan to recruit approx.15, 000 subjects for each city (average. 5,000 subjects for each community), and 120,000 subjects in total then comprise the national study sample. The plan will be updated, based on the prevalence obtained in the pilot study.

   1.3. Screening and diagnosis The screening tool will be chosen from Autism Spectrum Rating Scale (ASRS) or SRS（Social Responsiveness Scale） after pilot study.The questionnaire is a parent-administered form that takes approximately 15-20 minutes to complete. Parents of recruied children were invited to complete the questionnaire. Parents of all questionnaire screen-positive children will be contacted for appointing further diagnostic evaluations. Children whose parents could not be reached are classified as non-responders. The DSM-Ⅳ, ADI-R and ADOS (ADI-R: Autism Diagnosis Interview-Revised, ADOS: Autism Diagnosis Observation Scales) are used for diagnostic evaluations. Co-morbidities, such as epilepsy and ADHD (Attention Deficit Hyperactivity Disorder )after aditional medical examinations such as, EEG(electroencephalogram), head circumference, anthropometrics, allergies, sleep patterns, etc.
2. Risk Factors study on ASD A classic case-control design is applied to explore the risk factors of ASD. 2.1. Study subjects 2.1.1. Cases and control Cases were children living in target communities who are identified as positive based on questionnaire screen and the subsequent diagnosis with DSM-Ⅳ, ADOS and ADI-R.

Controls were children who are screened to be negative and matched to cases by age, gender, and class.

2.2. Environmental pollutants exposures Given the hypothesis that environmental factors might play a role in the etiology of ASD, we will analyze the biological samples of the subjects to investigate environmental exposures including chronic lead exposure, pesticides exposure, and endocrine disruptors exposure , for which, hair, blood, and urine will be collected for cases and controls. The detailed protocol for the measurement of each kind of biological sample has been introduced everywhere (see the references in individual block).

2.3. Analysis of other potential risk factors This study will also analyze the association between the onset of ASD and other risk factors, including diet (), living environment(),perinatal characteristics of parents, feeding history, baby growth and development after birth by using questionnaire and reviewing medical records.

2.4. Genetic analysis We are going to use the targeted area capture technology developed before and HiSeq2000, the second generation of high throughput sequencing platform, to carry out the molecular diagnosis screening (monogenic disease). Also, we will screen through Trio those ASD-related genetic mutations that are of high credibility and occur frequently so as to classify ASDs according to their definite etiologies.Furthermore, we will continue the study on the distribution of ASD relevant gene mutations among patients in China, which will lay a solid foundation for further studies of molecular epidemiology.Meanwhile, we will also apply genome-wide sequencing technology on the positive cases so as to find new mutation that might serve as potential molecular markers facilitating the diagnosis and treatment of ASDs.

A pilot study involving 4 cities (n=400 for each, in total n>=1600)will be conducted to test all methodology that will be applied in the prevalence study. A diagnostic study will be performed to evalute the performance of ASRS and SRS in screening ASD, one of which will be applied in the main study.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 6-12 years old and have lived in the recruied community over 6 months.

Exclusion Criteria:

* None

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community-based populations aged 6-12 years old form 8 cities in China
Sampling Method: Non-Probability Sample
Enrollment: 143755 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
prevalence of autism spectrum disorder | 3-12 years
  The outcome of the study include ASD and its commorbidities. The disease occurs in children as early as 18 months old, however the confirmation of diagnosis usually is 3 or later. 6-12 years is time frame for confirmed diagnosis.

SECONDARY OUTCOMES:
ASRS | 6-18 years
  ASRS is a measure for screen ASD.
ADI-R | 4-18 yeas
  The ADI-R is a good diagnosis tool for children with ASD
ADOS | 14months-16 years
  The ADOS is a appropriate instrutment for ASD diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Wang, PhD,MD, Principal Investigator — Children's Hospital of Fudan University
Locations (8):
- China (8):
  - Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Third Affiliated Hosptial,Sun Yat-Sen University, Guangzhou, Guangdong
  - Harbin Medical University, Harbin, Heilongjiang
  - Central South University, Changsha, Hunan
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Sichuan University, Chengdu, Sichuan
  - The 2nd Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Yan W, Siegert RJ, Zhou H, Zou X, Wu L, Luo X, Li T, Huang Y, Guan H, Chen X, Mao M, Xia K, Zhang L, Li E, Li C, Zhang X, Zhou Y, Shih A, Fombonne E, Zheng Y, Han J, Sun Z, Jiang YH, Wang Y. Psychometric properties of the Chinese Parent Version of the Autism Spectrum Rating Scale: Rasch analysis. Autism. 2021 Oct;25(7):1872-1884. doi: 10.1177/13623613211004054. Epub 2021 Apr 12. PMID 33845648
- [Derived] Zhou H, Zhang L, Wu L, Zou X, Luo X, Xia K, Wang Y, Xu X, Ge X, Sun C, Deng H, Fombonne E, Jiang YH, Yan W, Wang Y. Validity and reliability analysis of the Chinese parent version of the Autism Spectrum Rating Scale (6-18 years). Psychiatry Res. 2015 Dec 15;230(2):255-61. doi: 10.1016/j.psychres.2015.09.003. Epub 2015 Sep 8. PMID 26384573
- See also: The Children's Hospital of Fudan University (CHFU) is a service of the National Institute on Children — http://ch.shmu.edu.cn/